CLINICAL TRIAL: NCT07231666
Title: Goldilocks' Zone: Optimised Osmolality in Supplements for the Patient With an Ileostomy
Brief Title: Optimised Osmolality in Oral Supplements Optimised Osmolality in Oral Supplements
Acronym: Goldilocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1-10-72-289-21
Record Dates: First submitted 2022-08-01; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ileostomy - Stoma; Intestinal Failure
Keywords: Ileostomy; osmolality; natriuresis; dehydration; electrolyte
MeSH Terms: conditions — Intestinal Failure; Dehydration | interventions — Water; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: This was a single-centre, quasi-randomised cross-over intervention study. The effects of osmolality in oral supplements were investigated using a 3x3 cross-over design.
Who Masked: Participant
Masking Description: The patients were randomised to receive either the hypo-osmolar or hyper-osmolar in their first intervention. Microsoft Excel feature "RAND" (Microsoft version 16) was used to randomize oral supplements. Each supplement was assigned a number. Every time a patient agreed to one or two more intervention periods, two supplements were randomized. One of the primary investigators (JQ) enrolled and randomized supplements to the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hypoosmolar (Active Comparator): One with a hypo-osmolar fluid
  Interventions: Dietary Supplement: water
- isoosmolar (Active Comparator): one with an iso-osmolar fluid
  Interventions: Dietary Supplement: semi skimmed milk or powerade
- hyperosmolar (Active Comparator): one with a hyper-osmolar
  Interventions: Dietary Supplement: juice

INTERVENTIONS:
Dietary Supplement: water — oral commercially available supplements
  Arms: hypoosmolar
Dietary Supplement: semi skimmed milk or powerade — oral commercially available supplements
  Arms: isoosmolar
Dietary Supplement: juice — oral commercially available supplements
  Arms: hyperosmolar

SUMMARY:
Quasi-randomized, crossover intervention study, testing osmolality in oral drinks and effect on 6-hours ileostomy output in adult patients with an ileostomy

DETAILED DESCRIPTION:
14 patients with ileostomies were included in a quasi-randomized, crossover intervention study. Each patient ingested between 3-18 different supplements during separate 6-hours intervention periods. Ileostomy output and urine volume will be collected. Outcome measures include faecal wet-weight, urine volume, electrolytes, osmolality, and body composition measured with bioelectrical impedance analysis.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or higher
2. ileostomy formed at least 8 weeks before enrolment
3. consent to participate

Exclusion Criteria:

1. pregnancy
2. known chronic kidney disease
3. known diabetes mellitus
4. too long driving distance
5. parenteral nutrition/fluid more than 6 litres per month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
ileostomy output | 6 hours
  ileostomy output (wet weight feces grams)

SECONDARY OUTCOMES:
natriuresis | 6 hours
  urine volume (mL)
urine sodium | 6 hours
  urine sodium mmol
urine osmolality | 6 hours
  urine osmolality (mmol/kg)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of medicine V (Hepatology and Gastroenterology), Aarhus C
  - Aarhus University Hospital, Aarhus N

REFERENCES:
- [Result] Quist JR, Rud CL, Frumer K, Julsgaard M, Dahl Baunwall SM, Hvas CL. Osmolality in oral supplements drives ileostomy output: Defining the Goldilocks zone. Clin Nutr ESPEN. 2024 Jun;61:88-93. doi: 10.1016/j.clnesp.2024.03.003. Epub 2024 Mar 15. PMID 38777478